

Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

**Detailed Title:** An epidemiology study to assess *Plasmodium falciparum* 

parasite prevalence and malaria control measures in catchment areas of two studies pre- and post RTS,S/AS introduction (EPI-MAL-002 and EPI-MAL-003) to assess, in field conditions, vaccine benefit:risk in children in sub-

Saharan Africa.

SAP Version: Amendment 2 Final

**SAP Date:** *08APR2020* 

**Scope:** All data pertaining to the above study

GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, ppD



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

#### **TABLE OF CONTENTS**

| | | | PAGE |
|-----|--------------|--------------------------------------------------|------|
| LIS | ST OF A | ABBREVIATIONS | 4 |
| 1. | DOCU | JMENT HISTORY | 5 |
| 2. | STUD | OY DESIGN | 6 |
| | 2.1. | Study design overview | |
| | 2.2. | Study groups | |
| 3. | OBJE | CTIVES | 10 |
| | 3.1. | Co-Primary objectives | 10 |
| | 3.2. | Secondary objectives | |
| | 3.3. | Tertiary objectives | 10 |
| 4. | | POINTS | |
| | 4.1. | Primary endpoints | |
| | 4.2. | Secondary endpoints | |
| | 4.3. | Tertiary endpoints | 12 |
| 5. | STUD | Y POPULATION | 12 |
| 6. | STATI | ISTICAL METHODS | 13 |
| | 6.1. | Demography, medical history and fever | |
| | 6.2. | Analysis of parasite prevalence | |
| | 6.3. | Analysis of Malaria control interventions | |
| | 6.4.<br>6.5. | Analysis of parasite prevalence trends | |
| | 0.5. | 6.5.1. Microscopy | |
| | | 6.5.1.1 Descriptive analysis | |
| | | 6.5.1.2. Comparison analysis | |
| | | 6.5.2. NAAT results | |
| | | 6.5.2.1. Descriptive analysis | |
| | | 6.5.2.2. Comparison analysis | |
| | 0.0 | 6.5.3. Comparison between microscopy and NAA | |
| | 6.6. | Vaccination history | |
| | 6.7.<br>6.8. | Change in care seeking behaviours | |
| | 6.9. | Geographical heterogeneity Malaria risk factors | |
| | 6.10. | Malaria control programme at centre level | |
| | 6.11. | Analysis of SAEs related to study procedure | |
| | 6.12. | Output dataset | |
| 7. | STATI | ISTICAL CALCULATIONS | 10 |
| • | 7.1. | Methodology for computing CI | |



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

| | 7.2. | Number | of decimals | 3 | 19 |
|---|---|---|---|---|---|
| | 7.3. | Handling | missing da | ata | 19 |
| | 7.4. | Derived | and transfo | ormed data | 19 |
| | | 7.4.1. | Age | | 19 |
| | | | | Age at vaccination | |
| | | 7.4.2. | Definition | of vaccine eligible/ineligible age group | 20 |
| | | 7.4.3. | | of RTS,S/ AS01 <sub>E</sub> vaccination status | |
| | | 7.4.4. | | of a subject infected by a parasite – Slide | |
| | | | reading pa | arasitemia results at subject level | 21 |
| | | | 7.4.4.1. | Microscopy | 21 |
| | | | 7.4.4.2. | NAAT | 22 |
| | | 7.4.5. | Parasite p | revalence | 22 |
| | | 7.4.6. | | he study visit | |
| | | 7.4.7. | Other med | dication | 22 |
| | | 7.4.8. | Vaccination | on | 22 |
| | 7.5. | Prevaler | nce over all | sites | 23 |
| | 7.6. | Modellin | g of risk fac | ctors and malaria control interventions | 23 |
| | 7.7. | <b>Parasite</b> | mia prevale | ence trends | 24 |
| | 7.8. | | | | |
| | 7.9. | Rapid D | iagnostic Te | est (RDT) | 25 |
| | 7.10. | Malaria | risk factors | adaptation | 25 |
| 8. | COND | UCT OF | ANALYSES | S | 25 |
| | 8.1. | | | ses | |
| | 8.2. | • | • | ations for interim analyses | |
| 9. | CHAN | GES FRO | OM PLANNI | ED ANALYSES | 27 |
| 10 | REFE | RENCES | | | 27 |
| | | 1000 | | | |

Form Owner: VVHS Biometrics, PPD



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

The SAP is divided into 2 parts:

- first part detailing the analyses to be performed (current document)
- second part: annexe (called TFL) describing the flow and format of tables, figures and listings to be annexed to the SR.

### LIST OF ABBREVIATIONS

**ACT** Artemisinin-based combination therapy

**ATP** According to protocol Confidence interval CI **CTRS** Clinical Trial Registry Electronic case report form **eCRF** Generalized estimating equations **GEE** 

GlaxoSmithKline **GSK** Informed consent form **ICF** 

**IPTi** Intermittent preventative treatment in infants

Indoor residual spray **IRS** 

**JTEG** Joint technical expert group

LLLower limit

**LSAF** Life Science Analytics Framework Nucleic acid amplification test **NAAT** 

OR Odds Ratio

P. falciparum Plasmodium falciparum

P. vivax, P. Plasmodium vivax, Plasmodium malariae, Plasmodium Ovale

malariae, P. ovale

Personally identifiable information PII

Quantitative nucleic acid sequence-based amplification **QT-NASBA** 

Quantitative polymerase chain reaction **QT-PCR** 

Rapid diagnostic test **RDT** 

**RTS** Hybrid protein comprising HBs (hepatitis B surface antibody)

and CSP portions

Particulate antigen, containing both RTS and HBs proteins RTS.S

**SAE** Serious adverse event SAP Statistical Analysis Plan **SAR** Statistical Analysis Report

SD Standard Deviation

Seasonal malaria chemoprevention **SMC** Tables, Figures and Listings **TFL** 

Upper limit UL

World Health Organization **WHO** 

FORM-9000026972-01 Statistical Analysis Plan Template

Effective date: 08APR2020

GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, PPD

01June2014




Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

### 1. DOCUMENT HISTORY

| Date | Version | Description |
|---|---|---|
| 22-SEP-2015 | Final | |
| 19-DEC-2016 | Amendment 1 | <ul> <li>Cohen's Kappa coefficient added for the comparison between microscopy and NAAT (tertiary objective)</li> <li>Precisions added regarding the age derivation</li> <li>Update following protocol amendment 1 (from 5 surveys to 9 surveys)</li> </ul> |
| 08-APR-2020 | Amendment 2 | <ul> <li>Update following protocol amendment 2: <ul> <li>The study is extended from 9 surveys to 10 surveys</li> <li>Changes in sites participating according to sites enrolled in EPI-MAL-002 and EPI-MAL-003 studies.</li> <li>Update the definition of vaccine eligible/ineligible subgroup based on assumptions on the duration of the EPI-MAL-005 study and dates of RTS,S vaccine implementation start.</li> </ul> </li> <li>Update of computation rules to manage discrepancies detected during the first surveys and already mentioned in previous SAR.</li> <li>Additional analyses to support the EPI-MAL-003 study analysis and interpretation.</li> <ul> <li>Demographic tables and endpoints from primary objectives will be analysed by gender, JTEG age group, vaccine eligible group and RTS,S vaccine group.</li> <li>Adaptation of the trends analysis due to the update of the sites and the extension of the study.</li> <li>Details of the dataset that will be incorporated into analyses from EPI-MAL-002 and EPI-MAL-003 studies are removed and will be further detailed in their respective SAPs.</li> </ul> </ul> |

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* 

GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, PPD



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

#### 2. STUDY DESIGN

### 2.1. Study design overview

- Type of design: A multi-centric, epidemiology longitudinal cross-sectional study at centres in sub-Saharan Africa that are participating in GSK's EPI-MAL-002 and EPI-MAL-003 studies.
- There will be no study vaccine administered in this epidemiology study.
- Study population: Subjects 6 months to <10 years of age.
- Type of study: self-contained
- All medications that may influence malaria parasitaemia within 14 days prior to each survey will be recorded.
- Axillary body temperature of all subjects at the time of the survey will be recorded.
- Biological Samples: A capillary blood sample will be obtained for evaluation of malaria infection by blood slide and NAAT. In the event of measured fever at the time of the visit (axillary temperature ≥37.5°C) or fever reported in the last 24 hours or other symptoms/signs of clinical malaria, a rapid diagnostic test (RDT) will be conducted. If the RDT is positive, treatment will be given according to National guidelines. If a subject for whom no RDT was required is identified as being parasite positive following microscopy, National guidelines should be followed for clinical management of the subject.
- Microscopy and NAAT will be used to evaluate the level of asexual and sexual parasitaemia.
- Serious adverse events (SAEs) associated with the study procedure (capillary blood sampling) will be collected.
- Using Geographic Information System (GIS) to determine geographical variability in MTI locally: Study areas will be mapped by villages using grid referencing. Subjects will be attributed to their village, however, to avoid PII (personally identifiable information), small villages will be grouped when the number of participants is less than 10, so that it is not possible to identify one subject from one village. Therefore the study area will be divided into segments with a minimum of 10 subjects by segment regrouping villages by proximity if needed. Villages will be grouped at the time of random sampling of the study population. A map will be drawn showing the location of numbered segments, each numbered with a unique ID code and containing one or more villages. This map will NOT be submitted to GSK, but segments will be reported by their ID code and surface (km²) and subjects will be attributed to a segment code in the study database.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* GSK SOP Reference: SOP-9000026972



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

- Each study site will be requested annually to provide centre specific information about interventions from the malaria control program in the study area and, if facilities are available, to provide meteorological data for the study site such as rainfall and temperature. The information will be collected in the form of a questionnaire that will be recorded in a separate database to that for subject-specific data.
- Data collection: Electronic Case Report Form (eCRF).
- This study will involve up to 10 annual cross-sectional surveys during malaria peak transmission with possible further extension, dependent on the duration of the EPI-MAL-002 and EPI-MAL-003 studies.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* 

GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, ppD



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

#### 2.2. **Study groups**

The following group names will be used for the statistical analyses:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| P. falciparum infection status measured by microscopy | | |
| 1 | PF_INF | Subjects infected by P. falciparum parasitemia* |
| 2 | NOT_INF | Subjects not infected by P. falciparum parasitemia |
| 3 | UNK | Unknown |
| P. falciparum infe | ction status measured b | by NAAT |
| 1 | PF_INF_NAAT | Subjects infected by <i>P. falciparum</i> parasitemia* |
| 2 | NOT_INF_NAAT | Subjects not infected by P. falciparum parasitemia |
| 3 | UNK_NAAT | Unknown |
| Age classes acco | ording JTEG definition [y | ears] |
| 1 | 0.5-4Y | 6 months – 4 years at ICF date |
| 2 | 5-9Y | 5 – 9 years at ICF date |
| 3 | UNK | Unknown |
| Age classes acco | ording WHO definition [y | ears] |
| 1 | 0.5-1Y | 6 months – 1 year at ICF date |
| 2 | 2-9Y | 2 – 9 years at ICF date |
| 3 | UNK | Unknown |
| Vaccine eligible a | nge group | |
| 1 | Eligible | Vaccine eligible age group* |
| 2 | Ineligible | Vaccine ineligible age group* |
| RTS,S/AS01 <sub>E</sub> vac | ccination status | |
| 1 | Vaccinated | Children vaccinated with RTS,S/AS01 <sub>E</sub> malaria vaccine* |
| 2 | Unvaccinated | Children unvaccinated with RTS,S/AS01 <sub>E</sub> malaria vaccine* |
| Parasites density group measured by microscopy | | |
| 1 | Low | Low : < 2500 parasites/ µl |
| 2 | Medium | Medium : 2500 – 9999 parasites/ µl |
| 3 | High | High : 10000 – 19999 parasites/ μl |
| 4 | Vhigh | Very high : >= 20000 parasites/ µl |
| 5 | Neg | Negative |
| Parasites density group measured by NAAT | | |
| 1 | Low_NAAT | Low : < 1000 parasites/ µl |
| 2 | Medium_NAAT | Medium : 1000 – 10000 parasites/ μl |
| 3 | High_NAAT | High : > 10000 parasites/ µl |
| 5 | Neg_NAAT | Negative |

<sup>\*</sup> see section 7.4

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: 08APR2020

Form Owner: VVHS Biometrics, PPD

GSK SOP Reference: SOP-9000026972



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

Tables will, in general, be displayed by centre according to *P. falciparum* infection status and age classes. When it will not be the case (e.g. for some demographic tables), it will be explicitly mentioned.

According to the sites finally participating in the EPI-MAL-002 and EPI-MAL-003 studies, the following study sites names will be used for the statistical analyses:

| Site n° | Vaccine<br>exposed<br>status | Group label used in tables | Country | Districts (eCRF denomination - Demography) |
|---|---|---|---|---|
| Study site | Study site | | | |
| 207078 | Unexposed | 207078_BF_Nouna | Burkina<br>Faso | Nouna |
| 207079 | Unexposed | 207079_BF_Sapone | Burkina<br>Faso | Sapone |
| 207083 | Exposed | 207083_GH_Kintampo_EXP | Ghana | Kintampo North, Kintampo South,<br>Nkoranza North and Techiman North |
| 207083 | Unexposed | 207083_GH_Kintampo_UNEXP | Ghana | Nkoranza South and Techiman South |
| 228607 | Exposed | 228607_GH_Navrongo_EXP | Ghana | Kassena-Nankana West and East |
| 228607 | Unexposed | 228607_GH_Navrongo_UNEXP | Ghana | Builsa North and South |
| 235578 | Exposed | 235578_KE_Gem | Kenya | Gem (Siaya) |
| 235578 | Unexposed | 235578_KE_Bondo | Kenya | Bondo (Siaya) |
| 207082 | Exposed | 207082_KE_Kombewa | Kenya | Kombewa |
| 235579 | Unexposed | 235579_KE_Nyando | Kenya | Nyando |
| 233149 | Exposed | 233149_MA_Mangochi | Malawi | Exposed Malawi 1 |
| 233149 | Unexposed | 233149_MA_Monkey Bay | Malawi | Unexposed Malawi 1 |
| 233150 | Exposed | 233150_MA_St Monfort | Malawi | Exposed Malawi 2 |
| 233150 | Unexposed | 233150_MA_Chikwawa | Malawi | Unexposed Malawi 2 |
| 207080 | Unexposed | 207080_SN_Niakhar | Senegal | Niakhar |
| 207084 | Unexposed | 207084_SN_Keur Soce | Senegal | Keur Soce |
| 207081 | Unexposed | 207081_TZ_Korogwe | Tanzania | Korogwe |

The Senegal and Tanzania sites for which participation in the study was early terminated, were included in Survey 1 and Survey 2 only.

The Burkina Faso sites for which participation in the study was early terminated, were included in Survey 1 to Survey 4 only.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* 

GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, PPD



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

#### 3. OBJECTIVES

As per protocol.

### 3.1. Co-Primary objectives

In subjects aged  $\geq 6$  months and  $\leq 10$  years:

- To obtain longitudinal estimates of *P. falciparum* parasite prevalence in order to characterise malaria transmission intensity in a standardised way at centres conducting the EPI-MAL-002 and EPI-MAL-003 studies before and after the introduction of the malaria vaccine RTS,S/AS01<sub>E</sub> in sub-Saharan Africa.
- To obtain longitudinal estimates of the use of malaria control interventions in centres conducting the EPI-MAL-002 and EPI-MAL-003 studies before and after the introduction of the malaria vaccine RTS,S/AS01<sub>E</sub> in sub-Saharan Africa.

### 3.2. Secondary objectives

In subjects aged  $\geq 6$  months and  $\leq 10$  years:

- To estimate trends in longitudinal estimates of the parasite prevalence of *P*. *falciparum* by vaccine eligible or ineligible subgroups and overall.
- To obtain longitudinal estimates of the prevalence of *Plasmodium* species other than *P. falciparum*; overall and by age group.
- To estimate longitudinal trends in receipt and timing of the third dose of DTP/ HepB/Hib and the first dose of measles EPI vaccines, at around 14 weeks and 9 months of age respectively, as appropriate by country.
- To describe changes in care seeking behaviours for reported fever or malaria in the previous 14 days.
- To assess within-site geographical heterogeneity in malaria transmission intensity.
- To describe individual malaria prevention measures and risk factors for clinical malaria according to the parasite density observed.

### 3.3. Tertiary objectives

In subjects aged  $\geq 6$  months and  $\leq 10$  years:

- To compare asexual and sexual (gametocyte) parasitaemia (qualitative- and quantitative-density) in the RTS,S/AS01<sub>E</sub> vaccinated and unvaccinated subjects.
- To compare asexual and sexual gametocyte parasitaemia (qualitative- and semi-quantitative-density) when measured by microscopy or NAAT.

Effective date: 08APR2020 GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, ppp

FORM-9000026972-01 Statistical Analysis Plan Template



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

#### 4. ENDPOINTS

As per protocol.

### 4.1. Primary endpoints

• Occurrence of *P. falciparum* parasitaemia (using microscopy).

Criteria/definitions: infection determined using a blood smear slide and determined using microscopy.

• Occurrence of malaria control interventions.

Criteria/definitions: malaria control measures are mosquito net usage (including insecticide-treated nets [ITN] and long-lasting insecticidal nets [LLIN]), indoor, residual spraying (IRS), seasonal malaria chemoprevention (SMC), intermittent preventative treatment in infants (IPTi), and ACT therapy received within the last 14 days.

### 4.2. Secondary endpoints

Demography and history characteristics

Criteria/definitions: gender, age, medical history.

• Occurrence of *Plasmodium* species other than *P. falciparum* (using microscopy)

Criteria/definitions: infection with *Plasmodium* species other than *P. falciparum* determined using a blood smear slide and microscopy.

• Occurrence of uptake and timing of the third dose of DTP/HepB/Hib and the first measles EPI vaccines

Criteria/definitions: vaccination record of receipt of dose 3 of the DTP/HepB/Hib and the first dose of the measles EPI vaccines.

Occurrence of anti-malarial therapy

Criteria/definitions: any anti-malarial therapy received in the last 14 days.

Occurrence of measured fever

Criteria/definitions: any measured fever at time of visit (axillary temperature  $\geq$ 37.5°C).

Occurrence of reported fever

Criteria/definitions: any reported fever occurring in the last 24 hours.

01June2014 



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

Occurrence of care seeking behaviour

Criteria/definitions: occurrence of visits to health providers following reported fever or malaria in the previous 14 days.

Geo-referencing characteristics

Criteria/definitions: positioning of the subject's residence will be attributed to a segment with a unique ID from the grid referencing study area map in which the subject resides, where necessary, grouping small geographically proximate villages so that each segment has at least 10 study subjects to avoid PII, and proceeding as far as geographically appropriate.

• Occurrence of individual malaria prevention measures and risk factors

Criteria/definitions: malaria prevention measures are repellents and local herbs not specifically recommended by the national programme and risk factors are rural/urban area, construction material for the house, floor and roof, type of eaves (open/closed), use of electricity and water source (distance from and type).

### 4.3. Tertiary endpoints

Occurrence of RTS,S/AS01<sub>E</sub> vaccine doses

Criteria/definitions: vaccination record of each dose received of the RTS,S/AS01<sub>E</sub> vaccine.

• Occurrence of *P. falciparum* parasitaemia (using NAAT)

Criteria/definitions: detection of *P. falciparum* on dried blood spot and determined using NAAT.

• Occurrence of *P. falciparum* parasitaemia (using microscopy)

Criteria/definitions: detection of *P. falciparum* using a blood smear slide and determined using microscopy.

• Occurrence of sexual *P. falciparum* (using NAAT/QT-NASBA)

Criteria/definitions: detection of *P. falciparum* on dried blood spot and determined using NAAT.

#### 5. STUDY POPULATION

As per protocol.

As a reminder, the Total cohort will include all subjects enrolled in the study. All the information for these subjects will be collected in the eCRF (after receiving signed informed consent).

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, PPD



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

The According to Protocol (ATP) cohort will include all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures defined in the protocol, with no elimination criteria during the study) for whom at least one laboratory result of the blood sample is available.

A detailed, comprehensive list of reasons for elimination from ATP analyses will be established at the time of data cleaning and the following elimination codes will be used.

| Cohort | Elimination codes | Eli Type* |
|---|---|---|
| Total cohort | 900 | MA |
| ATP cohort | 2010 (inclusion/exclusion criteria) and 2500 (no slides reading available) | MA |

<sup>\*</sup>Internal GSK database code for type of elimination code

#### 6. STATISTICAL METHODS

As per protocol. SAS version 9.2 or above will be used for statistical analysis.

Continuous variables will be described with number of non-missing observations, mean, standard deviation (SD), median, minimum and maximum and number of missing observations. Categorical variables will be described with frequency tables; absolute numbers and percentages for each level will be given. For some categorical variables 95% confidence intervals (CIs) will also be presented.

All the analyses concerning objectives will be performed on the ATP cohort.

The analysis will be done also on the Total cohort only if we have more than 5% of eliminated subjects; except for the demography where all the tables will be performed for both cohorts.

### 6.1. Demography, medical history and fever

The number of subjects enrolled as well as the number excluded from the ATP analysis will be presented.

The distribution of subjects by centre will be tabulated according to *P. falciparum* infection status *measured by microscopy* and by both JTEG and WHO age classification.

Demographic characteristics (age at Informed Consent date, gender, previous enrolment) will be summarized by *P. falciparum* infection status *measured by microscopy* and overall, according to vaccine eligible status (see section 7.4.2) and RTS,S/AS01<sub>E</sub> vaccination status (see section 7.4.3 – only for the surveys starting after the introduction of the vaccine), using descriptive statistics.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* GSK SOP Reference: SOP-9000026972

GSK SOP Reference: SOP-900002697 Form Owner: VVHS Biometrics, PPD



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

Fever in the last 24 hours, fever at the visit, antimalarial or any other medication taken in the past 14 days will be tabulated by centre, and overall according to *P. falciparum* infection status and parasite density *measured by microscopy*.

### 6.2. Analysis of parasite prevalence

The analysis of co-primary objective regarding the *P. falciparum* parasitemia prevalence (defined in section 7.4.5) will be done for each centre separately and by age group (WHO and JTEG) and annual age, according to vaccine eligible status (see section 7.4.2), or RTS,S/AS01<sub>E</sub> vaccination status (see section 7.4.3 – only for the surveys starting after the introduction of the vaccine) *and by gender*. The pooled prevalence estimate will be computed considering the centre as random effect (as detailed in section 7.5). The heterogeneity among centres will be tested using Cochran's Q test based upon inverse variance weights.

This analysis of prevalence will be performed on the ATP cohort.

### 6.3. Analysis of Malaria control interventions

The bednet history information (sleeping under a mosquito net night before visit, new net, pierced or impregnated bednet, and how many holes) will be tabulated by centre, and overall according to *P. falciparum* infection status and parasite density *measured by microscopy*, *gender*, *vaccine eligible status* (see section 7.4.2), RTS,S/AS01<sub>E</sub> vaccination status (see section 7.4.3 – only for the surveys starting after the introduction of the vaccine) and JTEG age group.

The analysis of co-primary objective regarding the use of malaria control interventions will be done by computing the proportions of subjects using malaria control interventions among the subjects for which this information is available by centre and overall according to *P. falciparum* infection status and parasite density *measured by microscopy* and according to *gender*, vaccine eligible status (see section 7.4.2), *RTS*,*S*/*AS01*<sub>E</sub> vaccination status (see section 7.4.3 – only for the surveys starting after the introduction of the vaccine) and JTEG age group.

The CIs will be computed using the exact method.

Odds Ratio (OR) (unadjusted and adjusted) will be computed (see section 7.6).

This analysis will be performed on the ATP cohort

### 6.4. Analysis of parasite prevalence trends

The analysis of trends of parasitemia prevalence *measured by microscopy* (defined in section 7.7) will be performed only for the final analysis (i.e. at the last cross sectional-

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: **08APR2020** 

01June2014

GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, ppp



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

surveys), and in the ATP cohort. It will be done for each centre separately and according to vaccine eligible status (see section 7.4.2).

We will compute the *P. falciparum* parasitemia prevalence (defined in section 7.4.5) for each centre separately by survey year. And the pooled prevalence estimate will be computed considering the centre as random effect (as detailed in section 7.5).

Graphs will be performed to summarize the *P. falciparum* parasitemia prevalence according to vaccine eligible status (see section 7.4.2) and survey year, by centre.

### 6.5. Slide reading results

The analysis of slide readings (availability of slide readings, Malaria RDT results, slide methodology used, filter paper collection, number of days between date of slide reading and collection date) will be performed on the ATP cohort and will be done at the subject level (as defined in section 7.4.4) overall and by centre according to P. falciparum infection status measured by microscopy.

#### 6.5.1. Microscopy

#### 6.5.1.1. Descriptive analysis

The analyses of *P. falciparum* and gametocytes will be performed using descriptive statistics for each centre separately and overall and according vaccine eligible status (see section 7.4.2) and RTS,S/AS01<sub>E</sub> vaccination status (see section 7.4.3 – only for the surveys starting after the introduction of the vaccine). The density of *P. falciparum* parasitemia and gametocytes will also be evaluated.

The analyses regarding the prevalence of *Plasmodium* species other than *P. falciparum* will be done according to *P. falciparum* infection status measured by microscopy and vaccine eligible status (*see section 7.4.2*).

The distribution of *P. falciparum* and density measured by microscopy (with CIs) will be summarized for each centre separately and overall according to bednet use, and according to fever at the visit.

The results of *P. falciparum* and density measured by microscopy will also be computed according to the gametocytes results and the malaria RDT.

#### 6.5.1.2. Comparison analysis

The Fisher exact test will be used to perform the comparison, by RTS,S/AS01<sub>E</sub> vaccination status, of *P. falciparum* results measured by microscopy (see section 7.8).

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, PPD



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

#### 6.5.2. NAAT results

#### 6.5.2.1. Descriptive analysis

The analyses of *P. falciparum* and gametocytes will be performed using descriptive statistics for each centre separately and overall and according to vaccine eligible status (see section 7.4.2) and RTS,S/AS01<sub>E</sub> vaccination status (see section 7.4.3 – only for the surveys starting after the introduction of the vaccine).

The results of *P. falciparum measured by NAAT* will also be computed according to the gametocytes results *measured by NAAT*.

#### 6.5.2.2. Comparison analysis

The Fisher exact test will be used to perform the comparison, by RTS,S/AS01<sub>E</sub> vaccination status, of *P. falciparum* results measured by NAAT (see section 7.8).

#### 6.5.3. Comparison between microscopy and NAAT

The comparison of the *P. falciparum results and density* and gametocytes results measured by microscopy and by NAAT will be performed using the Cohen's Kappa coefficient [Cohen, 1960].

Simple Kappa coefficient will be used to compare the 2x2 contingency tables for the qualitative results (Positive/Negative, see section 7.4.4 for the details of categories).

For semi-quantitative results (see section 7.4.4 for the details of categories), simple and weighted Kappa coefficients will be used to compare the 4x4 contingency tables. The categories High: 10000 - 19999 parasites/  $\mu$ l and Very high:  $\ge 20000$  parasites/  $\mu$ l for the *microscopy* results will be pooled for this analysis.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* 

GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, PPD



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

The extent of the concordance will be assessed using the Landis and Koch scale [Landis, 1977]:

| Kappa | Interpretation |
|-----------|--------------------------|
| 0-0.20 | Slight agreement |
| 0.21-0.40 | Fair agreement |
| 0.41-0.60 | Moderate agreement |
| 0.61-0.80 | Substantial agreement |
| 0.81-1 | Almost perfect agreement |

### 6.6. Vaccination history

The vaccination history (which vaccine and age at vaccination) about DTP, Pentavalent, Measles and RTS,S/AS01<sub>E</sub> will be summarized overall and by *P. falciparum* infection status *measured by microscopy* using descriptive statistics.

### 6.7. Change in care seeking behaviours

The malaria or fever treatment taken in the past 14 days and details (where, when and at what time was the subject taken for treatment), and the malaria hospitalization will be displayed by centre, and overall according to P. falciparum infection status measured by microscopy.

### 6.8. Geographical heterogeneity

The distribution of subjects by segment will be tabulated according to *P. falciparum* infection status *measured by microscopy*.

Characteristics of segment will be summarized overall using descriptive statistics.

The analysis the *P. falciparum* parasitemia prevalence *measured by microscopy* (defined in section 7.4.5) will be done for each segment separately according to the centre. The heterogeneity among segment by centre will be tested using Cochran's Q test based upon inverse variance weights.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, PPD



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

#### 6.9. Malaria risk factors

The analysis of malaria risk factors will be performed on the ATP cohort.

The output tables for malaria risk factors (number of subjects in the same house, localisation, house information) will be done by centre and overall according to P. falciparum infection status and parasite density measured by microscopy. OR will be computed (see section 7.6).

#### 6.10. Malaria control programme at centre level

The centre specific data regarding the malaria control program will be summarized in the data listings by centre and by survey.

#### 6.11. Analysis of SAEs related to study procedure

SAEs reported during the entire study will be tabulated per centre and overall according to P. falciparum infection status measured by microscopy for the Total cohort.

#### 6.12. **Output dataset**

Annual fluctuations in malaria incidence occur as a result of changes in transmission intensity, which may be caused by changes in environmental factors such as rainfall or changes in usage of other malaria control interventions (use of bednets for example). Therefore, by taking into account these variations in MTI and malaria control intervention coverage, more accurate estimations of the vaccine impact on malaria disease diagnosed by RDT and/or microscopy during EPI-MAL-003 will be possible. Those estimations will be used as covariates in the models, as described in the protocol of the EPI-MAL-003.

EPI-MAL-005 is planned to run in parallel with EPI-MAL-002 and EPI-MAL-003 and will assess the following parameters: prevalence of *P. falciparum* parasitaemia, use of malaria control interventions, changes in environmental factors such as rainfall, changes in health care seeking behaviour, within-site geographical heterogeneity in MTI and individual malaria prevention measures and risk factors for malaria. Compliance with DTP-based, measles and RTS,S/AS01<sub>E</sub> vaccines will also be collected.

In order to adjust the comparison, and the estimation of the vaccine impact, an output dataset of the EPI-MAL-005 results will be built so that they could be included as covariates in the EPI-MAL-003 and EPI-MAL-002 models. This dataset will consist of aggregated results by centre, and by survey. These aggregated results will be explicitly listed in the appendices of the SAP of the EPI-MAL-003 and Epi-MAL-002 studies with the explanation of the models used.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: 08APR2020 GSK SOP Reference: SOP-9000026972

Form Owner: VVHS Biometrics, PPD



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

#### 7. STATISTICAL CALCULATIONS

### 7.1. Methodology for computing CI

All CI will be two sided 95% CI.

The exact 95% CIs for a proportion within a group will be calculated from Proc StatXact [Clopper, 1934].

The asymptotic 95% CIs for a mean within a group will be calculated.

#### 7.2. Number of decimals

The following decimal description will be used for the analyses.

| Parameters | Number of decimal digits |
|-------------------------------------|---------------------------------------|
| % of count, including LL & UL of CI | 1 |
| p-value | 4 |
| Minimum, maximum, range | Number of decimals in the raw data |
| Mean, median | Number of decimals in the raw data +1 |
| SD | Number of decimals in the raw data +2 |

LL = Lower Limit UL = Upper Limit CI = Confidence Interval

### 7.3. Handling missing data

No data handling will be performed in case of missing data.

#### 7.4. Derived and transformed data

#### 7.4.1. Age

The age will be computed as the difference between the informed consent date and the date of birth or taken directly as reported in the CRF if the date of birth is unavailable. The age will be categorized according to the JTEG definition: 0.5-4, 5-9 years and WHO definition: 0.5-1, 2-9 years.

When the age is derived from the informed consent date and the date of birth, it could be possible that the date of birth will not be a full date. When the date will be only a year, it will be read as "30JUNyyyy" (except for the year of the survey – given that it is known per inclusion criteria the subject is at least 6 months old). When the date will be a month and a year, it will be read as "15mmmyyyy". For these cases, the minimum age of the infant must be 6 months.

The continuous variable 'Age at IC [years]' is computed based on number of days/365.25.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: **08APR2020** 

GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, ppp

SD = Standard deviation



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

#### 7.4.1.1. Age at vaccination

The age at vaccination will be computed as the difference between the vaccination date and the date of birth.

It could be possible that the date of vaccination will not be a full date. When the date will be a month and a year, it will be read as "15mmmyyyy" except if the age becomes negative or is equal to zero, in which the date of birth will be used. When the date of vaccination will be only a year, the age at vaccination will not be derived.

If 3 different dates for the DTP/HepB/Hib vaccine are entered, the last date of vaccination is selected as the date of the third dose of DTP/HepB/Hib.

#### 7.4.2. Definition of vaccine eligible/ineligible age group

The vaccine eligible age group is defined as those subjects that on the basis of age would be eligible for RTS,S/AS01<sub>E</sub> vaccination, even if vaccine is unavailable at the time of assessment. The age will depend on the label for RTS.S/AS01<sub>F</sub> vaccination in the country. (At the time of study start, there will be no available vaccination with RTS,  $S/AS01_E$ ).

The vaccine ineligible age group is defined as those subjects that on the basis of age would be ineligible for RTS, S/AS01<sub>E</sub> vaccination, regardless of vaccine availability at the time of assessment. The age will depend on the label for RTS,S/AS01<sub>E</sub> vaccination in the country.

The cut-off age between both subgroups will be equal to the maximum age at *the last* survey for a child to be able to receive a RTS,S/AS01E vaccine dose.

After introduction of the RTS,S/AS01<sub>E</sub> vaccine in 2019 and based on Country MoH eligibility guidelines, the definition of vaccine eligible/ineligible group is defined as:

- RTS,S/AS01<sub>E</sub> vaccine ineligible group: regroup all subjects aged more or equal to 6 years except subjects who received at least one RTS,S vaccine dose.
- RTS, $S/AS01_E$  vaccine eligible group: regroup all subjects aged less than 6 years and the subjects aged more or equal to 6 years who received at least one RTS,S vaccine dose.

#### 7.4.3. Definition of RTS,S/ AS01<sub>E</sub> vaccination status

The vaccinated group is defined as those subjects who received at least one dose of the RTS, S/AS01<sub>E</sub> vaccine.

The unvaccinated group is defined as those subjects who received no dose of the RTS,S/AS01E vaccine.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: 08APR2020

01June2014

GSK SOP Reference: SOP-9000026972



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

The vaccination status will be determined only for the surveys/centres starting after the introduction of the vaccine.

Note: some vaccinated subjects were able to take part in clinical studies of the RTS,S/AS01<sub>E</sub> vaccine during phase III, so these subjects were vaccinated before the introduction of the vaccine.

# 7.4.4. Definition of a subject infected by a parasite – Slide reading parasitemia results at subject level

#### **7.4.4.1.** Microscopy

A subject is defined as infected by a specified parasite (*P. falciparum*, *P. malariae*, *P. vivax*, *P. ovale*) if at least two of his blood slide readings are positive for the corresponding parasite. Results of slide readings at subject level will be missing if all slide reading results are missing.

A subject is defined with presence of gametocytes when detected in at least one slide. It will be missing if all slide readings have missing information regarding the presence of Gametocytes.

The parasite density (parasites/µl) at the subject level is defined as the geometric mean of both (those positive) slide readings values if the subject's status is defined as positive. In the case of three positive slide readings, the two closest readings will be selected to calculate the geometric mean. In the case of negative parasite status, the density will be missing. If there are 3 values for one subject that have the same 'gap' between the lowest and the medium readings and between the medium and highest readings, the 2 greatest values (corresponding to the worst situation) are taken.

The parasites density will be categorized according to the following classes:

- Negative
- Low: < 2500 parasites/  $\mu$ l
- Medium : 2500 9999 parasites/ μl
- High: 10000 19999 parasites/ μl
- Very high :  $\geq$  20000 parasites/  $\mu$ l

For the concordances analyses the parasites density will be categorized according to the following classes:

- Negative
- Low: < 2500 parasites/  $\mu$ l

Form Owner: VVHS Biometrics, PPD

- Medium : 2500 9999 parasites/ μl
- High and Very high : >=10000 parasites/ μl

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* GSK SOP Reference: SOP-9000026972



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

The gametocytes density (units/ $\mu$ l) at the subject level is defined as the geometric mean of positive slide readings values if the subject status is defined as positive. It will be missing otherwise.

#### 7.4.4.2. NAAT

By the NAAT method, a subject is defined as infected by the *P. falciparum* or defined with presence of gametocytes if the NAAT reading is positive. Results of slide readings at subject level will be missing if the result is Not Done or Not Received.

The parasites density will be categorized according to the following classes:

- Negative
- Low :  $< 1000 \text{ parasites/ } \mu \text{l}$
- Medium : 1000 10000 parasites/ μl
- High: > 10000 parasites/  $\mu$ l

### 7.4.5. Parasite prevalence

The parasite prevalence will be estimated as the proportion of subjects infected divided by the number of subjects tested. These parasites will be estimated using microscopy testing (primary and secondary analyses) and using NAAT (tertiary analyses). The CIs will be computed using the exact method.

#### 7.4.6. Fever at the study visit

The status of fever at the study visit will be derived from the body temperature (axillary temperature). The value 'Yes' will be given if the temperature is  $\geq 37.5$ °C.

When the route of  $t^{\circ}$  is missing, it will be considered to be the axillary route. If the route is rectal (or tympanic with rectal conversion), then the conversion in axillary will be done, by subtracting  $0.5^{\circ}$ C ( $T^{\circ}$ \_Axil =  $T^{\circ}$ \_Rectal -0.5).

#### 7.4.7. Other medication

A variable 'Other medication over 14 days prior to study visit' will be derived from the eCRF if a subject was administered with a drug which was not reported as an antimalarial drug.

#### 7.4.8. Vaccination

The vaccines DTP, Tetravalent and Pentavalent will be regrouped in one category and called 'DTP/HepB/Hib' as for the EPI-MAL-002 study.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, ppp



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

The variable "Tradename of the vaccine" will be used to determine which vaccine is attributed to the subjects. As this variable is a free text variable, an excel file with the correct description of the vaccine was implemented by the epidemiologist.

#### 7.5. Prevalence over all sites

The proportion of occurrence of the *P. falciparum* parasitemia over all sites will be computed based on the proportions observed in each centre. Centres will be treated as clusters and the estimates (with 95%CI) will be computed using generalized estimating equations (GEE) in order to take the correlation between subjects from each study/country into account. The GEE will be fitted using the SAS procedure GENMOD [Boos, 1992) and Rotnitzky, 1990], assuming an exchangeable correlation matrix.

### 7.6. Modelling of risk factors and malaria control interventions



The potential risk factors and malaria control interventions collected will be considered.

The list of these variables can be found in the TFL. Note that some categories could be grouped at the time of the analysis in case of low representativeness.

A first table will summarise the effect of each risk factor and malaria control interventions individually on the proportion of positive episodes using unadjusted OR (with its 95% CI).

To describe the nature of the relationship between the dependent variable (probability of being P. falciparum positive **measured by microscopy**) and possible explanatory variables, a multiple logistic regression model will be used. Using the Backward selection strategy (with P-value of 0.05 to stay in the model – SLSTAY = 0.05) and the method of Maximum Likelihood to estimate the parameters, the final regression equation will identify the number of possible significant risk factors. Finally, the equation will be

$$Logit(P_i) = Log\left(\frac{P_i}{1 - P_i}\right) = \alpha + \sum_j \beta_j X_j$$

where

 $P_i$  = probability for a subject to be infected

 $X_i = \text{significant risk factors}$ 

FORM-9000026972-01 Statistical Analysis Plan Template

Effective date: 08APR2020

GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, ppD 01June2014




Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

A second table will give the details for the estimated coefficient, the adjusted OR, and the associated p-value *by using the variable site as cluster*.

The adjusted analysis will be done on one hand for risk factors and for malaria control interventions separately and on the other hand for all variables as a whole.

For the adjusted model, the variables depending on another variable will be adapted to avoid introducing missing values in the model:

- If the variable "Antimalarial or any other medication within 14 days prior the study visit" = No, then the value for the variables "Antimalarial drug" and "Other medication over 14 days prior the study visit" is assigned to No.
- If the variable "Indoor residual spray used in past 12 months to spray interior walls of this part of the house" = No, then the value for the variable "Use of indoor residual spray number of months age" = No Residual Spray.
- If the variable "subject sleep under a mosquito net last night" = No, then the value for the variables "new net (less than 1 year)" "Impregnated Bednet" and "Pierced/torn Bednet" = No Mosquito Net.
- If the variable "Pierced/torn Bednet" = No, then the value for the variable "Number of holes" = No Pierced Bednet.
- The categories of the variable "Use of indoor residual spray number of months ago" will be regrouped to:
  - 1-2 months
  - 3-4 months
  - > 4 months
  - No Residual Spray.

### 7.7. Parasitemia prevalence trends

To determine if a parasitemia prevalence trends may exist across the surveys, a Cochran-Armitage trend test is computed.

As some sites were early terminated during the study and others started after the RTS,S/AS01<sub>E</sub> vaccine introduction, the Cochran-Armitage trend test will be computed only on centres with results for at least 3 surveys.

The Cochran-Armitage test is a method of directing chi squared tests toward narrow alternatives. The test is sensitive to the linearity between response variable and experimental variables and detects trends. [Cochran, 1954, Armitage, 1955].

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, PPD



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

To compute the OR of Survey year according to vaccine eligible status (*see section 7.4.2*) and for each *site*, a simple logistic regression model will be used (see section 7.6).

The survey's reference category will be the first survey of the centre.

#### 7.8. Fisher exact test

The comparisons of proportions for categorical variables will be done with Exact Fisher test. The p-values less than 0.05 will be used as an indicator that a difference between the two groups compared may exist. However since p-values will not be adjusted for multiplicity comparisons, they will have to be interpreted with caution.

### 7.9. Rapid Diagnostic Test (RDT)

According to protocol, an RDT is performed when the subject has fever at the time of the visit (axillary temperature  $\geq 37.5^{\circ}C$ ) or fever reported in the last 24 hours or, after amendment 1 of the protocol, other symptoms/signs of clinical malaria. However, several protocol deviations were detected during the first surveys concerning the RDT use, i.e., some centres performed an RDT on non-eligible subjects. Due to this deviation, additional tables will be computed on the RDT results restricted to subjects with fever at first surveys and to subjects with fever or symptoms/signs of clinical malaria at surveys following amendment 1 of the protocol.

### 7.10. Malaria risk factors adaptation

An inconsistency was identified during the analysis of survey 2 between the 2 nested variables "What are the main types of windows in the house?" and "Are there nets on the main windows of the house?" (household questionnaire).

For most of the subjects living in a house with "no window", the category "Nets not present" was ticked for the nested variable describing net characteristics.

As a priori living in a house with "no window" could be considered as a protective factor when living in a house with "Nets not present" could be considered as a risk factor for malaria; the team decided to attribute to all subjects living in a house with 'No Window' the value 'Other' for the variable describing net characteristics.

#### 8. CONDUCT OF ANALYSES

### 8.1. Sequence of analyses

10 analyses will be performed with possible further extension, depending on the duration of the EPI-MAL-002 and EPI-MAL-003 studies.

Description Analysis ID TFL short title

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* 

01June2014



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

| | (LSAF sub-folder) | |
|---|---|---|
| Information collected in the first annual cross sectional | ANALYSIS_E1_02 | Cross Survey 1 |
| survey | | |
| Information collected in the second annual cross sectional | ANALYSIS_E1_03 | Cross Survey 2 |
| survey | | |
| Information collected in the third annual cross sectional | ANALYSIS_E1_04 | Cross Survey 3 |
| survey | | |
| Information collected in the fourth annual cross sectional | ANALYSIS_E1_05 | Cross Survey 4 |
| survey | | |
| Information collected in the fifth annual cross sectional | ANALYSIS_E1_07 | Cross Survey 5 |
| survey | | |
| Information collected in the sixth annual cross sectional | ANALYSIS_E1_08 | Cross Survey 6 |
| survey | | |
| Information collected in the seventh annual cross sectional | ANALYSIS_E1_09 | Cross Survey 7 |
| survey | | |
| Information collected in the eighth annual cross sectional | ANALYSIS_E1_10 | Cross Survey 8 |
| survey | | |
| Information collected in the ninth annual cross | ANALYSIS_E1_11 | Cross Survey 9 |
| sectional survey | | |
| Information collected in the <i>tenth</i> annual cross sectional | ANALYSIS_E1_01 | Cross Survey 10 and |
| survey and trend analysis over the <b>10</b> years. | | Trend analysis |
| Dataset on EPI-MAL-005 results used as covariates in | ANALYSIS_E1_12 | NA . |
| EPI-MAL-002 analyses | | |
| Dataset on EPI-MAL-005 results used as covariates in | ANALYSIS_E1_13 | NA . |
| EPI-MAL-003 analyses | | |

The analysis ID associated in Life Science Analytics Framework (LSAF) could be updated according the needs of the study.

The tables or graphs that will be performed only in the last survey are clearly identified in the TFL.

## 8.2. Statistical considerations for interim analyses

Not applicable

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* 

GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, PPD



Study alias & e-track number(s): 116682 (EPI-MALARIA-005 BOD AME)

#### 9. CHANGES FROM PLANNED ANALYSES



#### 10. REFERENCES

Armitage, P (1955). "Tests for Linear Trends in Proportions and Frequencies". Biometrics (International Biometric Society) 11 (3): 375–386.

Boos, D. On Generalized Score Tests. The American Statistician 1992; 46, 327–333.

Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika* 1934; 26: 404-413.

Cochran, WG (1954). "Some methods for strengthening the common chi-squared tests". Biometrics (International Biometric Society) 10 (4): 417–451.

Cohen J. A coefficient of agreement for nominal scales. Educ Psychol Meas. 1960;(20):27-46.

Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics.mars 1977;33(1):159-74.

Rotnitzky, A. and Jewell, N. P. Hypothesis Testing of Regression Parameters in Semiparametric Generalized Linear Models for Cluster Correlated Data. *Biometrika* 1990; 77, 485–497.

FORM-9000026972-01 Statistical Analysis Plan Template Effective date: *08APR2020* GSK SOP Reference: SOP-9000026972

GSK SOP Reference: SOP-9000026972 Form Owner: VVHS Biometrics, ppp